CLINICAL TRIAL: NCT03399370
Title: A Placebo-Controlled, Double-Blind, Randomized Trial to Evaluate the Effect of 300 mg of Inclisiran Sodium Given as Subcutaneous Injections in Subjects With Atherosclerotic Cardiovascular Disease (ASCVD) and Elevated Low-Density Lipoprotein Cholesterol (LDL-C)
Brief Title: Inclisiran for Participants With Atherosclerotic Cardiovascular Disease and Elevated Low-density Lipoprotein Cholesterol
Acronym: ORION-10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-PCS-17-04
Record Dates: First submitted 2018-01-03; First posted 2018-01-16 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: ASCVD; Elevated Cholesterol
Keywords: Inclisiran sodium; ASCVD; LDL-C
MeSH Terms: conditions — Hypercholesterolemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Inclisiran sodium 300 milligrams (mg) will be administered as a SC injection on Day 1, Day 90, then every 6 months.
  Interventions: Drug: Inclisiran Sodium
- Saline Solution (Placebo Comparator): Placebo will be administered as a SC injection of saline solution on Day 1, Day 90, then every 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran Sodium — Inclisiran is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis.
  Arms: Inclisiran
Drug: Placebo — Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
  Other Names: Saline Solution
  Arms: Saline Solution

SUMMARY:
This is a Phase III, placebo-controlled, double-blind, randomized study in participants with ASCVD and elevated LDL-C despite maximum tolerated dose of LDL-C lowering therapies to evaluate the efficacy, safety, and tolerability of subcutaneous (SC) inclisiran injection(s). The study will be a multicenter study in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years of age.
2. History of ASCVD (coronary heart disease [CHD], cardiovascular disease [CVD], or peripheral arterial disease [PAD]).
3. Serum LDL-C ≥1.8 millimole (mmol)/liter (L) (≥70 mg/dL).
4. Fasting triglyceride <4.52 mmol/L (<400 mg/dL) at screening.
5. Participants on statins should be receiving a maximally tolerated dose.
6. Participants not receiving statins must have documented evidence of intolerance to all doses of at least 2 different statins.
7. Subjects on lipid-lower therapies (such as a statin and/or ezetimibe) should be on a stable dose for ≥30 days before screening with no planned medication or dose change during study participation.

Exclusion Criteria:

1. New York Heart Association (NYHA) class IV heart failure.
2. Uncontrolled cardiac arrhythmia
3. Uncontrolled severe hypertension
4. Active liver disease
5. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least 2 methods of highly effective contraception (failure rate less than 1% per year) (for example, combined oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, or intrauterine device) for the entire duration of the study. Exemptions from this criterion:

   1. Women >2 years postmenopausal (defined as 1 year or longer since last menstrual period) and more than 55 years of age.
   2. Postmenopausal women (as defined above) and less than 55 years of age with a negative pregnancy test within 24 hours of randomization.
   3. Women who are surgically sterilized at least 3 months prior to enrollment.
6. Males who are unwilling to use an acceptable method of birth control during the entire study period (such as condom with spermicide).
7. Treatment with other investigational products or devices within 30 days or 5 half-lives of the screening visit, whichever is longer.
8. Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1561 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wright, MD, Principal Investigator — Mayo Clinic
Locations (145):
- United States (145):
  - Research Site 10001-015, Birmingham, Alabama
  - Research Site 10001-138, Foley, Alabama
  - Research Site 10001-113, Huntsville, Alabama
  - Research Site 10001-058, Mobile, Alabama
  - Research Site 10001-037, Montgomery, Alabama
  - Research Site 10001-076, Saraland, Alabama
  - Research Site 10001-013, Chandler, Arizona
  - Research Site 10001-077, Mesa, Arizona
  - Research Site 10001-136, Phoenix, Arizona
  - Research Site 10001-051, Surprise, Arizona
  - Research Site 10001-019, Tucson, Arizona
  - Research Site 10001-004, Tucson, Arizona
  - Research Site 10001-132, Tucson, Arizona
  - Research Site 10001-073, Beverly Hills, California
  - Research Site 10001-050, Canoga Park, California
  - Research Site 10001-011, Carlsbad, California
  - Research Site 10001-065, El Cajon, California
  - Research Site 10001-150, Los Angeles, California
  - Research Site 10001-043, Northridge, California
  - Research Site 10001-022, Northridge, California
  - Research Site 10001-033, Sacramento, California
  - Research Site 10001-105, San Ramon, California
  - Research Site 10001-008, Santa Rosa, California
  - Research Site 10001-153, Spring Valley, California
  - Research Site 10001-044, Torrance, California
  - Research Site 10001-047, Boca Raton, Florida
  - Research Site 10001-084, Clearwater, Florida
  - Research Site 10001-155, Clearwater, Florida
  - Research Site 10001-099, Clearwater, Florida
  - Research Site 10001-127, Daytona Beach, Florida
  - Research Site 10001-119, Fleming Island, Florida
  - Research Site 10001-070, Fort Lauderdale, Florida
  - Research Site 10001-067, Hialeah, Florida
  - Research Site 10001-139, Jacksonville, Florida
  - Research Site 10001-039, Jacksonville, Florida
  - Research Site 10001-098, Jacksonville, Florida
  - Research Site 10001-081, Miami, Florida
  - Research Site 10001-140, Miami, Florida
  - Research Site 10001-142, Miami, Florida
  - Research Site 10001-030, Miami, Florida
  - Research Site 10001-089, Miami, Florida
  - Research Site 10001-116, Miami, Florida
  - Research Site 10001-080, Miami Springs, Florida
  - Research Site 10001-027, Pembroke Pines, Florida
  - Research Site 10001-115, Pembroke Pines, Florida
  - Research Site 10001-048, Pembroke Pines, Florida
  - Research Site 10001-147, Pembroke Pines, Florida
  - Research Site 10001-003, Pinellas Park, Florida
  - Research Site 10001-104, Ponte Vedra, Florida
  - Research Site 10001-090, Saint Augustine, Florida
  - Research Site 10001-123, Sarasota, Florida
  - Research Site 10001-102, St. Petersburg, Florida
  - Research Site 10001-038, Tampa, Florida
  - Research Site 10001-143, Tampa, Florida
  - Research Site 10001-069, Atlanta, Georgia
  - Research Site 10001-137, Dunwoody, Georgia
  - Research Site 10001-092, Macon, Georgia
  - Research Site 10001-059, Arlington Heights, Illinois
  - Research Site 10001-158, Chicago, Illinois
  - Research Site 10001-035, Chicago, Illinois
  - Research Site 10001-036, Evanston, Illinois
  - Research Site 10001-082, Indianapolis, Indiana
  - Research Site 1001-020, Sellersburg, Indiana
  - Research Site 10001-040, Valparaiso, Indiana
  - Research Site 10001-074, West Des Moines, Iowa
  - Research Site 10001-028, Hutchinson, Kansas
  - Research Site 10001-125, Lexington, Kentucky
  - Research Site 10001-108, Lexington, Kentucky
  - Research Site 10001-107, Owensboro, Kentucky
  - Research Site 10001-144, Crowley, Louisiana
  - Research Site 10001-041, Lake Charles, Louisiana
  - Research Site 10001-101, Monroe, Louisiana
  - Research Site 10001-024, Flint, Michigan
  - Research Site 10001-095, Grandville, Michigan
  - Research Site 10001-078, Sterling Heights, Michigan
  - Research Site 10001-034, Troy, Michigan
  - Research Site 10001-018, Edina, Minnesota
  - Research Site 10001-056, Saint Paul, Minnesota
  - Research Site 10001-156, St Louis, Missouri
  - Research Site 10001-007, St Louis, Missouri
  - Research Site 10001-053, Omaha, Nebraska
  - Research Site 10001-021, Omaha, Nebraska
  - Research Site 10001-112, Las Vegas, Nevada
  - Research Site 10001-124, Las Vegas, Nevada
  - Research Site 10001-060, Bridgewater, New Jersey
  - Research Site 10001-055, Raritan, New Jersey
  - Research Site 10001-054, Albany, New York
  - Research Site 10001-122, Binghamton, New York
  - Research Site 10001-128, Endwell, New York
  - Research Site 10001-042, New Windsor, New York
  - Research Site 10001-129, Poughkeepsie, New York
  - Research Site 10001-110, Williamsville, New York
  - Research Site 10001-063, Cary, North Carolina
  - Research Site 10001-064, Greensboro, North Carolina
  - Research Site 10001-145, Mooresville, North Carolina
  - Research Site 10001-046, Shelby, North Carolina
  - Research Site 10001-016, Akron, Ohio
  - Research Site 10001-120, Cincinnati, Ohio
  - Research Site 10001-154, Cincinnati, Ohio
  - Research Site 10001-010, Cincinnati, Ohio
  - Research Site 10001-134, Cincinnati, Ohio
  - Research Site 10001-014, Columbus, Ohio
  - Research Site 10001-012, Columbus, Ohio
  - Research Site 10001-141, Dayton, Ohio
  - Research Site 10001-148, Marion, Ohio
  - Research Site 10001-017, Edmond, Oklahoma
  - Research Site 10001-109, Wyomissing, Pennsylvania
  - Research Site 10001-001, Anderson, South Carolina
  - Research Site 10001-006, Greer, South Carolina
  - Research Site 10001-075., Greer, South Carolina
  - Research Site 10001-111, Myrtle Beach, South Carolina
  - Research Site 10001-133, Pelzer, South Carolina
  - Research Site 10001-026, Spartanburg, South Carolina
  - Research Site 10001-103, Rapid City, South Dakota
  - Research Site 10001-146, Athens, Tennessee
  - Research Site 10001-130, Kingsport, Tennessee
  - Research Site 10001-118, Knoxville, Tennessee
  - Research Site 10001-100, Amarillo, Texas
  - Research Site 10001-087, Austin, Texas
  - Research Site 10001-117, Austin, Texas
  - Research Site 10001-009, Dallas, Texas
  - Research Site 10001-068, Edinburg, Texas
  - Research Site 10001-126, Fort Worth, Texas
  - Research Site 10001-031, Houston, Texas
  - Research Site 10001-088, Houston, Texas
  - Research Site 10001-091, Houston, Texas
  - Research Site 10001-061, Houston, Texas
  - Research Site 10001-032, Houston, Texas
  - Research Site 10001-025, Lubbock, Texas
  - Research Site 10001-057, New Braunfels, Texas
  - Research Site 10001-106, Powell, Texas
  - Research Site 10001-079, Round Rock, Texas
  - Research Site 10001-071, San Antonio, Texas
  - Research Site 10001-083, Schertz, Texas
  - Research Site 10001-149, Shavano Park, Texas
  - Research Site 10001-045, Tomball, Texas
  - Research Site 10001-005, Layton, Utah
  - Research Site 10001-002, Salt Lake City, Utah
  - Research Site 10001-052, Salt Lake City, Utah
  - Research Site 10001-093, Falls Church, Virginia
  - Research Site 10001-085, Manassas, Virginia
  - Research Site 10001-094, Midlothian, Virginia
  - Research Site 10001-023, Richmond, Virginia
  - Research Site 10001-029, Suffolk, Virginia
  - Research Site 10001-114, Tacoma, Washington

REFERENCES:
- [Derived] Dutta S, Shah R, Singhal S, Singh S, Piparva K, Katoch CDS. A systematic review and meta-analysis of tolerability, cardiac safety and efficacy of inclisiran for the therapy of hyperlipidemic patients. Expert Opin Drug Saf. 2024 Feb;23(2):187-198. doi: 10.1080/14740338.2023.2293201. Epub 2023 Dec 19. PMID 38063346
- [Derived] Ray KK, Wright RS. Plain language summary of results from ORION-10 and ORION-11: two studies to learn how well inclisiran works in people with high cholesterol. Future Cardiol. 2023 Mar;19(4):175-184. doi: 10.2217/fca-2022-0133. Epub 2023 Jun 6. PMID 37282500
- [Derived] Ray KK, Wright RS, Kallend D, Koenig W, Leiter LA, Raal FJ, Bisch JA, Richardson T, Jaros M, Wijngaard PLJ, Kastelein JJP; ORION-10 and ORION-11 Investigators. Two Phase 3 Trials of Inclisiran in Patients with Elevated LDL Cholesterol. N Engl J Med. 2020 Apr 16;382(16):1507-1519. doi: 10.1056/NEJMoa1912387. Epub 2020 Mar 18. PMID 32187462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inclisiran | Saline Solution
Started | 781 | 780
Completed | 721 | 694
Not Completed | 60 | 86

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo will be administered as a SC injection of saline solution on Day 1, Day 90, then every 6 months.
  Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Placebo | Total
Number analyzed (Participants) | 781 | 780 | 1561
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 297 | 333 | 630
  >=65 years | 484 | 447 | 931
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.90) | 65.7 (8.89) | 66.0 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 232 | 478
  Male | 535 | 548 | 1083
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 9 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 7 | 3 | 10
  Black or African American | 110 | 87 | 197
  White | 653 | 685 | 1338
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 781 | 780 | 1561

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Placebo: Placebo administered as a subcutaneous injection of sterile saline solution (0.9% sodium chloride in water for injection) on Day 1, Day 90, and then every 6 months.
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
percent change | -56.34 [-58.35 to -54.34] | 1.30 [-1.24 to 3.83]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority — LS Mean Difference (95% CI) from Placebo; p < .0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -57.64, 95% CI 2-sided [-60.86 to -54.43] — Represents the least squares mean difference from Placebo

2. Primary Outcome: Time-adjusted Percentage Change in LDL-C Levels From Baseline After Day 90 and up to Day 540
Description: Assessments performed at Baseline, Day 90, Day 540, time-adjusted percent change at Day 540 reported
Time Frame: Baseline, Day 90 to Day 540
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Inclisiran: Inclisiran sodium 300 milligrams (mg) (equivalent to 284 mg inclisiran) administered as a subcutaneous injection on Day 1, Day 90, and then every 6 months.
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 790
percent change | -51.27 [-53.00 to -49.54] | 2.51 [0.77 to 4.25]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority — LS Mean Difference (95% CI) from Placebo; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -53.78, 95% CI 2-sided [-56.23 to -51.33] — Represents the least squares mean difference from Placebo

3. Secondary Outcome: Absolute Change in LDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
mg/dL | -56.18 [-58.47 to -53.90] | -2.06 [-4.36 to 0.24]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority — LS Mean Difference (95% CI) from Placebo; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -54.12, 95% CI 2-sided [-57.37 to -50.88] — Represents the least squares mean difference from Placebo

4. Secondary Outcome: Time-adjusted Absolute Change in LDL-C From Baseline After Day 90 and up to Day 540
Description: Assessments performed at Baseline, Day 90, Day 540, time-adjusted percent change at Day 540 reported
Time Frame: Baseline, Day 90 to Day 540
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
mg/dL | -53.66 [-55.41 to -51.92] | -0.39 [-2.14 to 1.37]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -53.28, 95% CI 2-sided [-55.75 to -50.80] — Represents the least squares mean difference from Placebo

5. Secondary Outcome: Percentage Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
percent change | -69.78 [-73.88 to -65.67] | 13.52 [9.28 to 17.77]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -83.80, 95% CI 2-sided [-89.25 to -77.34] — Represents the least squares mean difference from Placebo

6. Secondary Outcome: Percentage Change in Total Cholesterol From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 781
percent change | -33.56 [-35.09 to -32.03] | -0.42 [-1.95 to 1.11]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -33.13, 95% CI 2-sided [-35.30 to -30.97] — Represents the least squares mean difference from Placebo

7. Secondary Outcome: Percentage Change in Apolipoprotein B (ApoB) From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
percent change | -44.81 [-46.52 to -43.10] | -1.72 [-3.46 to 0.02]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < .0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -43.09, 95% CI 2-sided [-45.50 to -40.67] — Represents the least squares mean difference from Placebo

8. Secondary Outcome: Percentage Change in Non-HDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 781 | 780
percent change | -47.41 [-49.44 to -45.38] | -0.05 [-2.08 to 1.99]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -47.36, 95% CI 2-sided [-50.25 to -44.47] — Represents the least squares mean difference from Placebo

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Inclisiran | Saline Solution
All-Cause Mortality (participants affected / at risk) | 12/781 | 11/778
Serious Adverse Events (participants affected / at risk) | 175/781 | 205/778
Other Adverse Events (participants affected / at risk) | 247/781 | 219/778
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=781) | Saline Solution (N=778)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 14 | 12
Angina pectoris (Cardiac disorders) | 6 | 7
Angina unstable (Cardiac disorders) | 4 | 10
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 10 | 8
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 7 | 20
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 15 | 22
Coronary artery occlusion (Cardiac disorders) | 1 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 3 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 6 | 6
Nodal arrythmia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 4
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Ectopic hyperthyroidism (Endocrine disorders) | 1 | 0
Ophthalmic vein thrombosis (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Larger intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 3
Chest pain (General disorders) | 2 | 3
Death (General disorders) | 2 | 1
Gait disturbance (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 10 | 9
Pyrexia (General disorders) | 1 | 0
Sensation of foreign body (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 0 | 1
Vascular stent restenosis (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Cavernous sinus thrombosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticultis (Infections and infestations) | 2 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 1
Localised infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 2
Osteomyelitis acute (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Periotinitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 9
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 4
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Cardiac contusion (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Chemical burn (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Occupational exposure to product (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural hawmorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myelodyplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Carotid artery disease (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 3 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 3
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 2
Demetia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 7 | 4
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 2 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal subdural haematoma (Nervous system disorders) | 0 | 1
Status migrainosus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=781) | Saline Solution (N=778)
Bronchitis (Infections and infestations) | 46 | 30
Diabetes mellitus (Metabolism and nutrition disorders) | 120 | 108
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 39
Hypertension (Vascular disorders) | 42 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT03399370/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03399370/SAP_001.pdf